CLINICAL TRIAL: NCT00481364
Title: Atorvastatin Treatment to Attenuate the Progression of Cardiovascular Disease: Prospective, Randomized, Controlled Study
Brief Title: Atorvastatin Treatment to Attenuate the Progression of Cardiovascular Disease in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ercan OK (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Ercan OK, professor, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-4.1/2
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Vascular Calcification; Atherosclerosis; Dyslipidemia; Inflammation
Keywords: hemodialysis; endothelial function; coronary artery calcification; atherosclerosis; statin
MeSH Terms: conditions — Vascular Calcification; Atherosclerosis; Dyslipidemias; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Statin (Active Comparator): Atorvastatin 40 mg/day
  Interventions: Drug: atorvastatin
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 40 mg/day
  Arms: Statin
Drug: placebo — 1 tb/day
  Arms: Placebo

SUMMARY:
This prospective, randomized, controlled study aims to investigate the effects of atorvastatin treatment in hemodialysis patients concerning progression of coronary artery calcification, progression of carotid artery intima-media thickness, endothelial function, and inflammation.

DETAILED DESCRIPTION:
The effects of statin treatment on coronary artery calcifications, carotid artery intima-media thickness, and endothelial functions have never been investigated in hemodialysis patients. Regarding inflammation, the present data in hemodialysis patients are derived from small studies with short follow-up.

We postulate that atorvastatin would reduce progression of coronary calcification and carotid artery intima-media thickness, decrease inflammation, and improve endothelial function.

In this prospective, controlled, randomized study, four hundred forty-six prevalent hemodialysis patients who meet inclusion and exclusion criteria will be randomized to atorvastatin (20 mg/day in first month; increased to 40 mg/day afterwards) and placebo arms (each arm consists of 223 patients), after completion of baseline investigations. Randomization will be performed with random permuted blocks and will be stratified according to dialysis center, age, sex, diabetic status, duration of dialysis, high flux dialyser use, and dialysate calcium level. Follow-up period will be twelve months.

It is estimated that 446 patients would provide 90% power with a two-sided, alpha error rate of 5%, of detecting a significant difference between treatment arms. Dropout rate is expected to be 20%, not to be replaced.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80 years
* on maintenance bicarbonate hemodialysis scheduled thrice weekly, at least 12 hours/week
* willingness to participate to the study with a written informed consent

Exclusion Criteria:

* to have serious life-limiting co-morbid situations, namely active malignancy, active infection, end-stage cardiac, pulmonary, or hepatic disease
* to be scheduled for living donor renal transplantation
* pregnancy or lactating
* history of coronary bypass grafting, acute myocardial infarction or unstable angina pectoris confirmed by angiography within three months of randomization
* presence of an absolute indication to use lipid lowering drug or an absolute contraindication for lipid lowering therapy according to investigator's opinion
* history of statin sensitivity or adverse reaction to statins
* receiving any lipid-lowering agents within three months of randomization
* uncontrolled hypothyroidism defined as TSH level higher than 1.5 times of upper limit
* receipt of any investigational drug within 30 days before randomization
* inability to tolerate oral medication or history of significant malabsorption
* treatment with steroids or immunosuppressive drugs
* alcohol abuse, drug abuse
* ALT and/or AST levels more than three times above the upper limit of normal or symptomatic hepatobiliary disease
* unexplained CK > 3 times the upper limit of the normal range
* inability to give informed consent because of mental incompetence or a psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
progression of coronary artery calcification score | one year
progression of carotid artery intima-media thickness | one year
changes in the level of hsCRP | one year

SECONDARY OUTCOMES:
changes in the endothelial function | one year
changes in the level of hsCRP | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Ok, MD, Principal Investigator — Ege University, Division of Nephrology
Locations (1):
- Ege University School of Medicine, Division of Nephrology, Bornova, İzmir, Turkey (Türkiye)